CLINICAL TRIAL: NCT05317819
Title: A Randomized, Double-Blind, Multi-Center Study of ADI-PEG 20 Versus Placebo in Subjects With High Arginine Level and Unresectable Hepatocellular Carcinoma
Brief Title: Study of ADI-PEG 20 Versus Placebo in Subjects With High Arginine Level and Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POLARIS2021-001
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma; Advanced Hepatocellular Carcinoma
Keywords: Unresectable Hepatocellular Carcinoma; Genotype; Arginine; Arginine Deiminase; ADI-PEG 20; pegargiminase
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ADI PEG20

STUDY DESIGN:
Intervention Model Description: To evaluate efficacy and safety of ADI-PEG 20 or Placebo in patients with high-arginine-phenotypic and HCC
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a randomized, double-blind trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: ADI-PEG 20 (Experimental): Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM)
  Interventions: Drug: ADI-PEG20
- Drug: Placebo (Placebo Comparator): Dose: 36 mg/m2 given weekly Route of Administration: Intramuscular (IM)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ADI-PEG20 — Treatment for hepatocellular carcinoma
  Other Names: pegargiminase
  Arms: Drug: ADI-PEG 20
Other: Placebo — Treatment for hepatocellular carcinoma
  Arms: Drug: Placebo

SUMMARY:
Evaluate efficacy and safety of ADI-PEG 20 in patients with high-argininephenotypic and HCC

DETAILED DESCRIPTION:
Safety will be evaluated by laboratory tests, vital sign measurements, physical examinations and subject medical history which will be performed to detect new abnormalities and any deterioration in pre-existing conditions.

Efficacy will be determined by overall survival, progression free survival, pharmacodynamics (peripheral blood arginine and citrulline levels) and immunogenicity (antibodies to ADI-PEG 20).

ELIGIBILITY:
Inclusion Criteria:

1. Prior diagnosis of HCC confirmed by radiology, histology, or cytology.
2. Prior treatment with at least 1 systemic agent for Child-Pugh A subjects. However, Child-Pugh B7 subjects without prior systemic treatment may be enrolled, if they are not eligible for any approved systemic therapies (e.g., due to financial factors).
3. Plasma arginine ≥ 78 μM at pre-screening visit.
4. Measurable disease using RECIST 1.1 (Appendix A). At least 1 measurable lesion must be present. Subjects who have received local-regional therapies are eligible, provided that they have either a target lesion which has not been treated with local therapy and/or the target lesion(s) within the field of the local regional therapy has shown an increase of ≥ 20% in size. Local-regional therapy must be completed at least 4 weeks prior to the baseline CT scan.
5. Child-Pugh (cirrhosis status) score class A-B7 (Appendix C).
6. Barcelona Cancer of the Liver (BCLC) stage C (Appendix B)
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment (Appendix D).
8. Expected survival of at least 3 months.
9. Age >18 years.
10. Fully recovered from prior surgery, radiation, or chemotherapy, and none within 2 weeks prior to week 1 visit. Liver biopsy for HCC confirmation is allowed.
11. Female subjects and male subjects must be asked to use appropriate contraception for both the male and female for the duration of the study and for 35 days after last dose of ADI-PEG 20/placebo. Male partners of female subjects and female partners of male subjects must agree to use two forms of contraception or agree to refrain from intercourse for the duration of the study if they are of childbearing potential. Females of childbearing potential must not be pregnant at the start of the study, and a serum human chorionic gonadotropin (HCG) pregnancy test must be negative before entry into the study. If positive HCG pregnancy test, further evaluation to rule out pregnancy must be performed according to GCP before this subject is deemed eligible. Females not of childbearing potential must be post-menopausal (defined as cessation of regular menstrual period for at least 12 months).
12. Informed consent must be obtained prior to study initiation.
13. No concurrent investigational studies are allowed.
14. Total bilirubin < 3.0 mg/dL and no evidence of bile obstruction.
15. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤5 x upper limit of normal range.
16. Serum albumin level ≥ 3.0 g/dl.
17. Prothrombin time (PT)-international normalized ratio (INR): PT <3 seconds above control or INR <1.7.
18. Absolute neutrophil count (ANC) >1,500/µL.
19. Platelets >50,000/µL.
20. Serum uric acid ≤ 8 mg/dL (with or without medication control).
21. Serum creatinine ≤ 1.5 x the upper limit of normal range, or, if serum creatinine >1.5 x the upper limit of normal range, then the creatinine clearance must be ≥ 40 mL/min.
22. Subjects with active hepatitis B or C on anti-viremic compounds may remain on such treatment, except for interferon.
23. Encephalopathy - none or mild (grade 1 or 2, by Child-Pugh classification); lactulose of other supportive care allowed.
24. Ascites - absent or slight (by Child-Pugh classification); diuretic therapy allowed.

Exclusion Criteria:

1. Candidate for potential curative therapies (i.e., resection or transplantation) or eligible for approved systemic therapies according to the labeling of such drugs.
2. Prior allograft transplantation including liver transplantation.
3. Subjects who have not fully recovered from toxicities associated with previous HCC loco-regional or systemic therapies, except for Grade 1 alopecia.
4. Serious infection requiring treatment with intravenous, systemically administered antibiotics at the time of study entrance, or an infection requiring systemic antibiotic therapy within 7 days prior to the first dose of study treatment.
5. Pregnancy or lactation.
6. Expected non-compliance.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association Class III or IV), cardiac arrhythmia, or psychiatric illness, social situations that would limit compliance with study requirements.
8. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present or in the opinion of the investigator will not affect patient outcome.
9. Subjects who had been treated with ADI-PEG 20 previously.
10. History of uncontrolled seizure disorder not related to underlying cancer.
11. Allergy to pegylated compounds.
12. Allergy to E. coli drug products (such as GMCSF).
13. Bleeding esophageal or gastric varices within the prior three months, except if banded or treated.
14. Uncontrolled ascites (defined as not easily controlled with diuretic treatment).
15. Having received any blood transfusion, blood component preparation, erythropoietin, albumin preparation, or granulocyte colony stimulating factors (G-CSF) within 7 days prior to screening laboratories or after screening laboratories have been obtained until week 1 visit.
16. Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 18 months
  Time from study enrollment to death

SECONDARY OUTCOMES:
Progression free survival | Approximately 18 months
  Time from study enrollment to progressive disease or death

CONTACTS AND LOCATIONS:
Overall Officials: John S Bomalaski, Study Director — Polaris Group
Locations (11):
- Taiwan (8):
  - Changhua Christian Hospital (CCH), Changhua
  - Ditmanson Medical Foundation Chiayi Christian Hospital (CYCH), Chiayi City
  - Chang Gung Medical Foundation-Chia-Yi (CGMF-CY), Chiayi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital (KMUH), Kaohsiung City
  - Chang Gung Medical Foundation-Kaohsiung(CGMF-KS), Kaohsiung City
  - Chi Mei Medical Center (CMMC-YK), Tainan
  - Chi Mei Hospital, Liouying (CMMC-LY), Tainan
  - Chang Gung Medical Foundation-Linkou (CGMF-LK), Taoyuan District
- Vietnam (3):
  - Bach Mai Hospital, Hanoi
  - K Hospital, Hà Nội
  - Hue Central Hospital, Huế